CLINICAL TRIAL: NCT04568187
Title: Clinical Efficacy of Fat Reduction on the Thigh of Korean Women Through Cryolipolysis
Brief Title: Cryolipolysis Induced Gluteal Fat Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonik Trade Company, Korea (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 01177787
Record Dates: First submitted 2020-05-19; First posted 2020-09-29 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Body Weight Changes
Keywords: fat; cryolipolysis; Women; femoral fat
MeSH Terms: conditions — Body Weight Changes; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Intervention Model Description: the sequential split-body trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- cryolipolysis machine on Left inner thigh (Active Comparator): Zeltiq machine as intervention procedure was carried out on left inner thigh (treated side) for 1 hour through cool sculpting procedure with CIF (Cooling Intensity Factor: -73 mW/cm2).
  Interventions: Device: zeltiq
- radiofrequency on right thigh (Sham Comparator): The radio frequency method was applied on right thigh (control side) as sham procedure for 30 minutes through 3000 Hz- amplitude modulated frequency at once.
  Interventions: Device: placebo

INTERVENTIONS:
Device: zeltiq — Zeltiq prototype device (Zeltiq Aesthetics, Pleasanton, CA) approved by FDA 2010
  Arms: cryolipolysis machine on Left inner thigh
Device: placebo — radiofrequency with 3000 Hz
  Arms: radiofrequency on right thigh

SUMMARY:
There was no difference in efficacy in removal of local fat on thigh by cryolipolysis through Zeltiq machine.

Cryolipolysis was found to be safe for 12 week clinical trial.

DETAILED DESCRIPTION:
this study is conducted to investigate the clinical efficacy and safety of cryolipolysis on fat removal of thigh through cryolipolysis.

Healthy premenopausal volunteered women had been conducted to assess their anthropometrical, social, and cardio-metabolic, and femoral fat amount by computer tomography, and adverse events at initial, 4 week, 12 week visit.

ELIGIBILITY:
Inclusion Criteria:

* pre-menopausal healthy women
* subjects with body mass index ≥ 18
* subjects with visible fat on both thigh
* subjects to understand and agree to this study protocol

Exclusion Criteria:

* subjects with cryoglobulinemia, cold urticaria, or paroxysmal cold hemogobulinemia
* subjects with pregnancy or lactation within 6 months or next 3 months
* subjects with any laboratory, or metabolic abnormalities
* uncooperative subjects to comply with the study protocol
* women taking any medication/ over the counter/herbal supplements to regulate weight or fat mass over 6 months
* subjects with menstrual irregularities
* subjects to change over 10% of the former weight within the past 6 months - any procedure such as liposuction, or another surgical procedure or mesotherapy to reduce fat within 6 months
* subjects with any dermatologic abnormalities on the target areas (thigh)
* subjects with any injection into the area of intended treatment (e.g. cortisone) within 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy Women
Enrollment: 15 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2010-08-31 (Actual)

PRIMARY OUTCOMES:
The change of girths in both thighs | 4 weeks
  Comparison of circumferences of both thighs
The change of fat amounts in both thighs | 4 weeks
  Comparison of cross-sectional areas in both thighs

SECONDARY OUTCOMES:
The change of girths in both thighs | 12 weeks
  Comparison of circumferences of both thighs
The change of fat amounts in both thighs | 12 weeks
  Comparison of cross-sectional areas in both thighs

CONTACTS AND LOCATIONS:
Overall Officials: Kyu R Lee, MD, PhD, Principal Investigator — Hongik General Hospital
Locations (1):
- Bariatric clinic/Family medicine, Hong-Ik General Hospital, Seoul, South Korea

REFERENCES:
- See also: clinical efficacy of fat reduction on the thigh of Korean women through cryolipolysis — http://dx.doi.org/10.4172/2165-7904.1000203